CLINICAL TRIAL: NCT04328584
Title: Intraoperative Navigation for Surgically Precise Resection of the Chest (INSPIRE)
Acronym: INSPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-6162
Record Dates: First submitted 2020-03-24; First posted 2020-03-31 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Thoracic Wall
MeSH Terms: interventions — Surgical Navigation Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SNS (Experimental): Intraoperative imaging/surgical navigation system (SNS)
  Interventions: Procedure: surgical navigation system

INTERVENTIONS:
Procedure: surgical navigation system — Navigation system providing surgeons with an additional view of the chest wall lesion

SUMMARY:
While undergoing chest wall resection, a surgeon's major concern is obtaining an appropriate surgical margin. Difficulty or failure to do so can result in prolonged operative time, need for re-operation due to a positive resection margin, or need for complex chest wall reconstruction due to unnecessarily wide resection. Over the last decades, surgical navigation systems have been developed to improve operative precision in various surgical fields. This is achieved by integrating patient images with intraoperative findings.

DETAILED DESCRIPTION:
Integration of CT imaging systems into the operating room now provide real-time 3D images of patient anatomy during surgery. This better adjusts for anatomical deformation and tissue excision compared to using preoperative images alone.

Twenty patients scheduled for chest wall resection will be enrolled over the study duration of 2 years. Patients will undergo imaging and surgery in the GTx-OR at Toronto General Hospital, as part of the GTx Program of the TECHNA Institute. All patients will be asked to consent to receiving their care in a research environment. They will also be asked to consent to having the intraoperative image acquired and used to generate a navigation view in the GTx-OR. Instead of resecting the chest wall lesion according to the preoperative images alone with intraoperative findings as per standard-care procedures, the navigation view will be used as an additional reference for surgeons during the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent
2. Scheduled to undergo surgical resection of a chest wall lesion
3. At least 18 years of age
4. Must sign and be given a copy of the written informed consent form

Exclusion Criteria:

1. Unresectable lesions or unstable patient condition, for which surgery is not recommended
2. Participants with metallic implantation, such as ribs fixations, a pacemaker, or pedicle screws, which may affect the accuracy of CBCT
3. Excluded at the discretion of the clinical investigator/surgeon, if they are enrolled in other studies that will result in combined radiation exposure exceeding standard of care
4. Pregnant, lactating, or planning to become pregnant during the period of the evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Performance metrics for navigation-assisted chest wall resection | 2 years

SECONDARY OUTCOMES:
Image accuracy metrics - Intraoperative CBCT and preoperative CT will be compared to confirm accuracy in predicting the anatomical relationship of lesions with adjacent structures. | 2 years
Incident reports of OR-related delays and malfunctions | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided